CLINICAL TRIAL: NCT01664572
Title: Methodological Issues of Laser Speckle Contrast Imaging for Studying Microcirculation.
Brief Title: Methodological Issues and Laser Speckle Contrast Imaging
Acronym: METHODO-LSCI
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2012A00458-35
Record Dates: First submitted 2012-08-07; First posted 2012-08-14 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Microvascular Function
Keywords: laser Doppler flowmetry, skin blood flow

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy subjects

SUMMARY:
Microcirculation, especially skin microcirculation, is a window towards systemic vascular function in magnitude and underlying mechanisms. Different techniques have been developed to assess the microcirculation. Among these techniques, laser technology is used to perform non-invasive microvascular assessments. Although this technique is widely used, different methodological issues remain. This study aims at defining the way to use lasers for clinical use.

ELIGIBILITY:
Inclusion Criteria:

* age > 18years old
* subject without any known cardiovascular disease

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of France
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2012-06; Primary Completion 2015-09 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Angers, France

REFERENCES:
- [Derived] Omarjee L, Signolet I, Humeau-Heutier A, Martin L, Henrion D, Abraham P. Optimisation of movement detection and artifact removal during laser speckle contrast imaging. Microvasc Res. 2015 Jan;97:75-80. doi: 10.1016/j.mvr.2014.09.005. Epub 2014 Sep 28. PMID 25261716
- [Derived] Puissant C, Abraham P, Durand S, Humeau-Heurtier A, Faure S, Leftheriotis G, Mahe G. Assessment of endothelial function by acetylcholine iontophoresis: impact of inter-electrode distance and electrical cutaneous resistance. Microvasc Res. 2014 May;93:114-8. doi: 10.1016/j.mvr.2014.04.001. Epub 2014 Apr 13. PMID 24735977
- [Derived] Puissant C, Abraham P, Durand S, Humeau-Heurtier A, Faure S, Leftheriotis G, Rousseau P, Mahe G. Reproducibility of non-invasive assessment of skin endothelial function using laser Doppler flowmetry and laser speckle contrast imaging. PLoS One. 2013 Apr 19;8(4):e61320. doi: 10.1371/journal.pone.0061320. Print 2013. PMID 23620742